CLINICAL TRIAL: NCT05027776
Title: Evaluating the Immunogenicity and Safety of Quadrivalent Human Papillomavirus Recombinant Vaccine (Type 6, 11, 16, 18) in Healthy Chinese Female Subjects Aged 9 to 26 Years: A Phase 3, Open-label, Non-randomized Clinical Trial
Brief Title: Immunogenicity and Safety of Quadrivalent HPV Vaccine in Healthy Chinese Female Subjects Aged 9 to 19 Years
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Bovax Biotechnology Co., Ltd. (Industry)
Collaborators: Chongqing Bovax Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-HPV-3002
Record Dates: First submitted 2021-08-20; First posted 2021-08-30 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: HPV Infections; Cervical Cancer Stage IIa; Vaginal Cancer; Genital Wart; CIN1; CIN2; CIN3
Keywords: Human papillomavirus; vaccine; Cervical Cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Vaginal Neoplasms; Condylomata Acuminata

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: 2-doses Group (Experimental): Subjects aged 9-14 years, received 2 doses of q-HPV vaccine, which was administered intramuscularly in the deltoid muscle of the non-dominant arm according to a 0, 6-month schedule.
  Interventions: Biological: 2-doses Group among 9-14 years
- Experimental: 3-doses Group (Experimental): Subjects aged 9-19 years, received 3 doses of q-HPV vaccine, which was administered intramuscularly in the deltoid muscle of the non-dominant arm according to a 0, 2，6-month schedule.
  Interventions: Biological: 3-doses Group among 9-19 years
- Acitve Group (Active Comparator): Subjects aged 20-26 years, received 3 doses of q-HPV vaccine, which was administered intramuscularly in the deltoid muscle of the non-dominant arm according to a 0, 2，6-month schedule.
  Interventions: Biological: 3-doses Group among 20-26 years

INTERVENTIONS:
Biological: 2-doses Group among 9-14 years — Subjects were planned to receive two doses of the study vaccine administered intramuscularly according to a 0, 6 month vaccination schedule.
  Arms: Experimental: 2-doses Group
Biological: 3-doses Group among 9-19 years — Subjects were planned to receive three doses of the study vaccine administered intramuscularly according to a 0, 2, 6 month vaccination schedule.
  Arms: Experimental: 3-doses Group
Biological: 3-doses Group among 20-26 years — Subjects were planned to receive three doses of the study vaccine administered intramuscularly according to a 0, 2, 6 month vaccination schedule.
  Arms: Acitve Group

SUMMARY:
This phase 3 study will evaluate the immunogenicity and safety of Quadrivalent HPV recombinant vaccine in Chinese females aged 9 to 26 years

DETAILED DESCRIPTION:
This is a singel-center study (protocol 4-HPV-3002) in which women are planned to receive q-HPV vaccine. Study participation will last approximately 60 months and involves a total of nine or eleven scheduled visits.

This study will also assess whether the immunogenicity of the q-HPV vaccine given 2-dose schedule in 9-14 year old girls is noninferior to that in young women, aged 20-26, receiving 3 doses, and 3 doses in 9-19 year old girls is noninferior to that in young women receiving 3 doses, while assessing the safety of this vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese females aged 9 to 26 years; Provide legal identification;
2. The subject voluntarily agrees to enroll in this study. If the subject is a minor, both the subject and subject's legal guardian should voluntarily agree to enroll in this study and sign an informed consent form;
3. Had a negative urine pregnancy test on the day of enrollment, among the subjects of childbearing age; Not in the duration of breast-feeding and no birth plan within 7 months; According to the investigator's judgment that there is no possibility of pregnancy at that time: subjects have taken effective contraception, or asexual life after the last menstrual period, or use IUD, or had undergone ligation; subjects agree to continue take effective contraception such as taking OCS and condom use;
4. No fever symptoms on the day of enrollment (aged> 14 years old, axillary temperature<37.3°C; aged ≤ 14 years old, axillary temperature<37.5°C );
5. Be able to understand the study procedures and promise to participate in regular follow-ups under the requirements;

Exclusion Criteria:

1. Received marketed HPV vaccine or plan to receive marketed HPV vaccine during this study period or have enrolled in HPV vaccine clinical trials;
2. Enrolling or plan to enroll in other clinical trials (drug or vaccine);
3. History of positive test to HPV, history of cervical cancer (e.g. abnormal screening test results, abnormal cervical biopsy results, including CIN, LSIL, and cervical cancer) or history of pelvic radiotherapyherpes;
4. History of diseases related to HPV infection (e.g. genital warts, VIN, VaIN, and related cancers) or history of STDs, including syphilis, gonorrhea, genital herpes, Mycoplasma genitalium, Lymphgranuloma Venereum, granuloma inguinale, etc.;
5. Known allergy to any vaccine components or history of severe allergic diseases requiring treatment, including shock, laryngeal edema, urticarial, Henoch-Schonlein purpura, Arthus reaction, etc.;
6. Had primary or acquired immunodeficiency such as HIV, SLE, JRA, etc;
7. History of epilepsy and convulsions (except fever convulsions in children under 5 years of age);
8. Subjects with existing infectious diseases such as TB, viral hepatitis, and/or HIV infection; or existing liver or kidney conditions, CVDs, and malignancy;
9. Untreated/uncontrolled hypertension before vaccination (aged 9 to 17 years: systolic BP≥120mmHg and/or diastolic BP≥80mmHg; aged more than 18 years: Systolic BP≥140mmHg and/or diastolic BP ≥90mmHg);
10. With prohibitive contraindications such as Thrombocytopenia or coagulopathy;
11. Asplenic, functionally asplenic, or splenectomy caused by any condition;
12. Received immunosuppressive treatment within one month before study such as long-term glucocorticoid use(≥2mg per kg per day, lasted more than two wks), or plan to receive such treatment from month 0 to month 7；
13. Receipt of immune globulin or blood-related products within 3 months; or plan to receive such products during this study period（month 0 to month 7）;
14. Within 3 days prior to vaccination, have an acute disease or are in the acute attack of a chronic disease or have used antipyretic, analgesic and anti-allergic drugs (such as: acetaminophen, ibuprofen, aspirin, loratadine, ceti Rizine, etc.);
15. Receipt of inactivated, RNA, and recombinant vaccines within 14 days, live vaccines within 28 days;
16. Subjects with existing mental illness, History of mental illness, or Family History;
17. According to the investigator's judgment, the subject has any condition may interfere with process of evaluation or participating in this study cannot guarantee the object's maximum benefit.

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1348 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Primary immunogenicity outcome | At month 8
  Number of subjects receiving the whole schedule vaccination with antibody responses as assessed by GMT and SCR, change from baseline among the seronegative vaccine recipients at Month 8

SECONDARY OUTCOMES:
Secondary immunogenicity outcome | At month 12, 24, 36, 48 and 60
  TNumber of subjects, aged 9 to 14, receiving the 2-doses scheduled vaccination with antibody responses as assessed by GMT and SCR, change from baseline among the seronegative vaccine recipients at Month 12, 24, 36, 48 and 60
Number of subjecs with AEs | Within 30 minutes (Days 0) after vaccination
  Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal, headache, myalgia, rash, fever (= axillary temperature above 37.3°C or 37.5°C) and urticaria.
Numbers of subjects with solication of AEs | Within 8 days (Days 0-8) after vaccination
  Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal, headache, myalgia, rash, fever (= axillary temperature above 37.3°C or 37.5°C) and urticaria.
Numbers of subjects with unsolicited AEs | Within days 0-30 after vaccination
  An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Number of subjects receiving the whole schedule vaccination with SAEs | Subjects receiving a 2-doses shceduled vaccination from Day o to Month 60; Subjects receiving a 3-doses shceduled vaccination from Day o to Month 12
  SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Number of subjects with pregnancy events | Subjects receiving a 2-doses shceduled vaccination from Day o to Month 60; Subjects receiving a 3-doses shceduled vaccination from Day o to Month 12
  Outcomes of pregnancies were Live infant NO apparent congenital anomaly (ACA) , Live infant, Elective termination NO ACA, Elective termination CA, Ectopic pregnancy, Spontaneous abortion NO ACA, Stillbirth NO ACA, Stillbirth CA, Lost to follow up and Pregnancy ongoing.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Huang, Study Director — Sichuan Provincial Center for Disease Control and Prevention
Locations (1):
- Center for Disease Control and Prevention, Mianyang, Sichuan, China